CLINICAL TRIAL: NCT01559038
Title: Canadian Humira Post Marketing Observational Epidemiological Study Assessing Effectiveness in Psoriatic Arthritis (Complete-PsA)
Brief Title: Canadian Humira Post Marketing Observational Epidemiological Study Assessing Effectiveness in Psoriatic Arthritis
Acronym: Complete-PsA
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Cato Research (Industry); JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-666
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2019-12

CONDITIONS: Psoriatic Arthritis
Keywords: Assessing Effectiveness in Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- adalimumab: Responding to treatment with non-biologic DMARDs (disease-modifying antirheumatic drugs) and initiated on treatment with adalimumab as monotherapy or in combination with other medications
- DMARD (disease-modifying antirheumatic drugs): Initiated on non-biologic DMARD(disease-modifying antirheumatic drugs) or requiring switching to another non biologic DMARD (disease-modifying antirheumatic drugs) as monotherapy, or in combination with other medications

SUMMARY:
The current study will assess the real - life effectiveness of adalimumab in the management of articular and dermatological manifestations of moderate to severe Psoriatic Arthritis (PsA).

ELIGIBILITY:
Inclusion Criteria:

* Adult >= 18 years old
* Has provided written informed consent allowing the use of their data for the study and providing permission for contact by the study personnel
* Active Psoriatic Arthritis (PsA) with three (3) or more tender and swollen joints as well as active psoriatic skin lesions or confirmed history of psoriasis
* Inadequate response or non-tolerant to current disease-modifying antirheumatic drugs (DMARD) based treatment for PsA

Exclusion Criteria:

* Currently participating in another prospective study including controlled clinical trials and observational studies
* Patient cannot or will not sign informed consent
* Stable disease with adequate tolerance and response to current treatment and no change in treatment is indicated
* Previous treatment with anti-tumor necrosis factor (anti-TNF) or other biologic agent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Offices of community rheumatologists & dermatologists
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2012-02-16 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Change in the Disease Activity Score - 28 (DAS-28) | Every 3 months up to 6 months, then every 6 months up to 24 months
  The DAS - 28 is calculated using the number of swollen (SJC) and tender (TJC) joints out of 28, the erythrocyte sedimentation rate (ESR) and the patient's global assessment of disease activity using a 100 mm visual analogue scale (VAS)

SECONDARY OUTCOMES:
Duration of Morning Stiffness (min) | Every 3 months up to 6 months, then every 6 months up to 24 months
  This is ascertained by the treating physician during the patient assessment and is measured in minutes
Dermatology Life Quality Index (DLQI) | Baseline, month 6, month12, month 24
  This is a self-administered questionnaire comprised of 10 items assessing a patient's skin and problems associated with skin disease. The 10 questions in the DLQI converge into six domains that measure symptoms and feelings, daily activities, leisure, work and / or school, personal relationships and satisfaction with treatment.
Health Assessment Questionnaire - Disability Index (HAQ-DI) | Every 3 months up to 6 months, then every 6 months up to 24 months
  Self-administered questionnaire measuring the patient's functional ability during the last week.
Patient Global Assessment of Disease Activity (VAS and 5 Point Scale) | Every 3 months up to 6 months, then every 6 months up to 24 months
  A 100 mm VAS with 0 indicating lowest disease and 100 highest disease activity and a five point Likert Scale (0 - 4) that is completed by the patient at the physician's office
Physician Global Assessment of Disease Activity (VAS and 5 Point Scale) | Every 3 months up to 6 months, then every 6 months up to 24 months
  This is a 100 mm VAS with 0 indicating lowest disease and 100 highest disease activity a five point Likert Scale (0 - 4) that is completed by the physician during the patient examination

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (41):
- Canada (41):
  - Pont, Cranbrook, BC, CA /ID# 69120, Cranbrook, British Columbia
  - Dr. Barbara T. Blumenauer Inc. /ID# 75393, Kamloops, British Columbia
  - Hudson, Kamloops, Canada /ID# 69104, Kamloops, British Columbia
  - Dr. Maqbool R. Sheriff Inc. /ID# 69125, Nanaimo, British Columbia
  - Carmi Medical Clinic /ID# 69128, Penticton, British Columbia
  - Dr. J. Antonio Avina-Zubieta /ID# 71035, Richmond, British Columbia
  - Dr. Alfonso Verdejo Inc. /ID# 69131, Vancouver, British Columbia
  - Dr. Milton F. Baker Inc. /ID# 69085, Victoria, British Columbia
  - Manitoba Clinic /ID# 69113, Winnipeg, Manitoba
  - Nexus Clinical Research /ID# 45622, St. John's, Newfoundland and Labrador
  - St. Clare's Mercy Hospital /ID# 69121, St. John's, Newfoundland and Labrador
  - Qe Ii Hsc /Id# 69129, Halifax, Nova Scotia
  - Dr. Juris Lazovskis Inc. /ID# 69111, Sydney, Nova Scotia
  - Waterside Clinique /ID# 72173, Barrie, Ontario
  - Shickh, Bowmanville, Canada /ID# 90513, Bowmanville, Ontario
  - Brockville Medical Center /ID# 69105, Brockville, Ontario
  - Dr. Sanjay Dixit Medicine Professional Corporation /ID# 69092, Burlington, Ontario
  - Dr. Chrisotomor Kouroukis & Dr /ID# 137894, Dundas, Ontario
  - Charlton Medical Centre /ID# 133073, Hamilton, Ontario
  - Charlton Medical Centre /ID# 69122, Hamilton, Ontario
  - Dr. William G. Bensen Centre /ID# 69086, Hamilton, Ontario
  - West Mountain Medical Center /ID# 128878, Hamilton, Ontario
  - Lynderm Research Inc. /ID# 76736, Markham, Ontario
  - Brandusa Florica Med Prof Corp /ID# 81876, Mississauga, Ontario
  - Credit Valley Rheumatology /ID# 69089, Mississauga, Ontario
  - Imtiaz MS Khan Medicine Prof /ID# 69110, Mississauga, Ontario
  - Rajwinder S. Dhillon Medicine /ID# 138672, Niagara Falls, Ontario
  - Davis, Ottawa, CA /ID# 69091, Ottawa, Ontario
  - Setty, Owen Sound, CA /ID# 69123, Owen Sound, Ontario
  - York Dermatology Clinic and Research Centre /ID# 127943, Richmond Hill, Ontario
  - Pedvis Med Prof Corp /ID# 69388, Toronto, Ontario
  - Jonathan Stein Med Prof Corp /ID# 71134, Toronto, Ontario
  - Karasik, Toronto, CA /ID# 69109, Toronto, Ontario
  - Institut de Rhum. de Montreal /ID# 69100, Montreal, Quebec
  - PSS Medical Inc. /ID# 69127, Montreal, Quebec
  - Couture, Outremont, CA /ID# 69090, Outremont, Quebec
  - Ctr. de Rheum de l'est du QC /ID# 69097, Rimouski, Quebec
  - Groupe de Recherche en Maladies Osseuses /ID# 69087, Sainte-Foy, Quebec
  - CHUS - Hopital Fleurimont /ID# 94735, Sherbrooke, Quebec
  - Ctr. de Recherche Musculo-Sque /ID# 69112, Trois-Rivières, Quebec
  - Rheum Disease Ctr of Montreal /ID# 143964, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khraishi MM, Remple VP, Silverberg S, Stewart JC, Florica B, Bessette L. Canadian Adalimumab Postmarketing Observational Epidemiological Study Assessing Effectiveness in Psoriatic Arthritis (COMPLETE-PsA): 12-month Results of Comparative Effectiveness of Adalimumab and nbDMARDs. J Rheumatol. 2022 May;49(5):454-464. doi: 10.3899/jrheum.200609. Epub 2022 Jan 15. PMID 35033999
- See also: Related Info — http://rxabbvie.com